CLINICAL TRIAL: NCT01294189
Title: The Impact of Instituting a Law for Advance Directives on End-of-life Decision Making in Intensive Care Medicine in Germany
Brief Title: Advance Directives and End-of-life Decision Making in Intensive Care Medicine in Germany
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Priv.-Doz. Dr. Jan-Peter Braun, Charite University, Berlin, Germany
Other Study IDs: EOLD
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-01

CONDITIONS: Death
Keywords: end-of-life decisions, critical care, advance directive
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- ICU-patients that died on the ICU: ICU-patients (post-operative and non operative patients) will be enrolled in the study. All patients are followed until their death on the ICU.

SUMMARY:
Description of the decision making process as well as the practices of end of life care in an ICU of a German university hospital during the period when changes of German legislation occurred.

DETAILED DESCRIPTION:
Most patients on the intensive care unit (ICU) die after an end-of-life decision (EOLD) has been made (Sprung et al. 2003). On September 1st 2009 the "advance-directives-law" was inured in Germany considering a written advance directive of an adult binding for physicians and the patient´s surrogate decision makers if it fits into the medical context (BGBL 2009). There is a lack of data describing the process and the factors associated with end-of-life-decisions in ICUs in Germany in detail.

The purpose of this observational study is to describe the decision making process as well as the practices of end of life care in an ICU of a German university hospital during a period when changes of German legislation occurred.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the ICU
* All patients discharged death from the ICU

Exclusion Criteria:

* All patients discharged alive from the ICU

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All intensive care department patients (MAN101i and MAN103i Charité Berlin) will be enrolled in the study
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2008-08; Primary Completion 2010-09 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
decision makers of end-of-life decisions | 08/2008 - 09/2010
  The primary objective of this study performed according to an observational post-ad-hoc design is to identify and analyse the decision makers of end-of-life decisions on an intensive care unit in Germany.
  Approximately 200 patients will be enrolled in the study. They are followed up until their death on the ICU. Usually in clinical routine end-of-life decisions are documented for decision makers in the patients´ records. The incidences of the different decision makers including members of different clinical specialities and also members with different levels of ICU experience are compared.

SECONDARY OUTCOMES:
influence of the new German advance directives law on end-of-life decisions | 08/2008 - 09/2010
  The second objective is to investigate what kind of influence the new German law for advance directives had on end-of-life decision making on the ICU.
  Approximately 200 patients will be enrolled in the study. They are followed up until their death on the ICU. Usually in clinical routine end-of-life decisions are documented for decision makers and procedures in the patients´ records. The incidences of therapeutic procedures in end of life care comparing patients with advance directives at different time points and those patients without advance directives are reviewed for differences.
the process of end-of-life decisions on a German intensive care unit | 08/2008 - 09/2010
  Another objective of this study performed according to an observational post-ad-hoc design is to identify and analyse the process of end-of-life decisions on an intensive care unit in Germany.
  Approximately 200 patients will be followed up until their death on the ICU. The process of withholding and withdrawing of therapeutic approaches is documented in the patient´s records. The incidences of different therapeutic procedures like ventilation, organ replacement technology, surgery, blood transfusions, antiinfective therapy and nutrition in patients with an EOLD are compared.

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Peter Braun, MD, Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine Campus Charité Mitte, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Graw JA, Spies CD, Wernecke KD, Braun JP. Managing end-of-life decision making in intensive care medicine--a perspective from Charite Hospital, Germany. PLoS One. 2012;7(10):e46446. doi: 10.1371/journal.pone.0046446. Epub 2012 Oct 1. PMID 23049701